CLINICAL TRIAL: NCT01813864
Title: Linking Services to Patient Needs for Improved Patient Outcomes (CASPAR)
Acronym: CASPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA015125 (NIH); 5R01DA015125-05 (NIH); NCT00797147 (obsolete NCT alias)
Record Dates: First submitted 2010-06-24; First posted 2013-03-19 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance Abuse
Keywords: treatment planning; resource guide; service matching; Service matching for substance abuse clients; CASPAR resource guide; Improved treatment planning
MeSH Terms: conditions — Substance-Related Disorders | interventions — casp protein, Drosophila; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CASPAR Resource Guide (Experimental): Treatment Enhanced/CASPAR-- All counselors in this study will receive a training and take part in the experimental arm of the study in Phase 2.
  Interventions: Behavioral: CASPAR/Treatment Planning

INTERVENTIONS:
Behavioral: CASPAR/Treatment Planning — All counselors in the study will receive additional training in treatment planning and the CASPAR Resource Guide software to easily identify and link patients to services not available at substance abuse treatment centers such as General Educational Development (GED) training, dental clinics, job training, etc.
  Other Names: CASPAR; Technology Tranfer; Assessment

SUMMARY:
The proposed Quality Improvement Initiative study is a health services research project in community-based substance abuse treatment programs. The primary goals are to use training and technology transfer to match services to client needs, increase the number of services received by clients, and improve client outcomes. This is a two phase study in which we compare clients pre-intervention to clients post-intervention.

Clients from Phase II (Post-Intervention) compared to Phase I (Pre-Intervention) will:have treatment plans that better match the problems reported at assessment; receive services that better match their needs, as reported during the assessment/intake; show better results during treatment performance on the Treatment Services Review (TSR), including attending a greater percentage of their scheduled treatment sessions and increased satisfaction with the Treatment Planning process; show better client outcomes at 3 month follow-up on primary drug and alcohol measures, including Breathalyzer and urine drug screen, and secondary personal health and social functioning measures such as days medical problems, days psychiatric problems, days employed, days of conflict with family members, etc.

DETAILED DESCRIPTION:
This protocol will specifically target identified organizational barriers by implementing the CASPAR system as a site-wide Quality Improvement Initiative (QI Initiative) study and enrolling seven sites in Bucks and Montgomery Counties in Pennsylvania and in the Southern New Jersey region who (1) were the most active sites in participating in the focus groups and provided feedback that led to the development of the new Quality Improvement protocol, (2) want to focus organizational effort and attention on improving treatment planning and problem-services matching, (3) met additional inclusion criteria (detailed below). They are all located within Bucks and Montgomery Counties in Pennsylvania and within a 70 mile radius of Atlantic City, New Jersey.

Executive directors at all invited programs will sign a Letter of Agreement (LoA) with Treatment Research Institute (TRI) that as an organization they will support their counselors in attending training, providing individualized treatment plans as well as monthly individualized sessions dedicated to problem-service matching; will add items necessary to their assessment to make sure it is equally comprehensive as the Addiction Severity Index (ASI), and will allow TRI to recruit clients for follow-up to evaluate the effectiveness of the QI Initiative implementation. The LoA will detail all site-specific expectations, along with benefits to the program, including free counselor and supervisor training (along with Certified Addictions Counselor (CAC) and Certified Alcohol Drug Counselor (CADC) credits), free software, and monetary compensation, $2,000 for site participation in Phase I of the study and $3,000 for site participation in Phase II of the study. Directors will also be provided with a detailed Director Information Sheet outlining aspects of the Quality Improvement Initiative outlined in the LoA.

TRI staff will provide counselors and supervisors with the treatment planning training as well as the CASPAR Resource Guide software and training on its use. These activities will be initiated as an organization-wide Quality Improvement Initiative, and as such, will be implemented with all counselors at each program. No data will be collected from the counselors, nor will we discuss or report on client outcomes grouped by counselor.

This will be a 2-Phase project. TRI staff will recruit up to 6 eligible clients per counselor prior to providing the CASPAR training and up to 6 additional clients after providing training. Based on current data from the sites, we expect a minimum of 36 counselors to be involved in the Quality Improvement Initiative.

Update June 1st 2009 - Based on current recruitment levels achieved and analysis needs, we are projecting recruitment of approximately 320 subjects.

We will continue to evaluate the effectiveness of this enhanced protocol by addressing the same aims and using primarily the same client instruments previously approved by this Institutional Review Board (IRB, some have been modified, see full discussion below). We will compare client outcomes before (Phase I) and after the individualized treatment planning and problem-service matching components are introduced (Phase II). As before, we expect to see pre-post differences in problem-treatment plan matching, treatment plan-service matching, and in the number and appropriateness of services clients receive; we also expect to see pre-post differences in client outcome such as treatment attendance, treatment retention, breathalyzer, and urinalysis results, the same measures and outcomes in the original design.

ELIGIBILITY:
Inclusion Criteria:

* currently attending substance abuse treatment

Exclusion Criteria:

* incarceration
* under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2004-08; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Better client outcomes at 3 month follow-up on primary drug and alcohol measures | 3 months post treatment start.

SECONDARY OUTCOMES:
Better client outcomes at 3 month follow-up on secondary personal health and social functioning measures such as days medical problems, days psychiatric problems, days employed, days of conflict with family members, etc. | 3-months post treatment start.
Increased satisfaction with the Treatment Planning process. | Assessed at 2, 4, 8 and 12 weeks.
Improved match between patient problems and treatment plan & services received. | Up to 3-months post treatment start.
  Improved match between:
  1. Patient problems identified at admission and treatment plan.
  2. Patient problems identified at admission and services received.

CONTACTS AND LOCATIONS:
Overall Officials: Deni Carise, PhD., Principal Investigator — Treatment Research Institute
Locations (7):
- United States (7):
  - SODAT, Camden, New Jersey
  - Cape Counseling, Cape May Court House, New Jersey
  - Genesis Counseling, Collingswood, New Jersey
  - SODAT, Woodbury, New Jersey
  - Aldie Counseling, Bensalem, Pennsylvania
  - Aldie Counseling, Doylestown, Pennsylvania
  - Malvern Institute, King of Prussia, Pennsylvania